CLINICAL TRIAL: NCT07256340
Title: Measuring Total Energy Expenditure in Critically Ill Patients Using the Doubly Labelled Water Method
Acronym: IC-TEE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/108
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: The study is a prospective, interventional trial with a single group design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DLW-based energy assessment (Experimental): Single-arm observational study
  Interventions: Diagnostic Test: DLW-based energy assessment

INTERVENTIONS:
Diagnostic Test: DLW-based energy assessment — Measuring TEE in IC patients with DLW

SUMMARY:
Critically ill patients, such as those with trauma or sepsis, experience high rates of malnutrition (up to 75%). Malnutrition worsens outcomes by increasing infection rates, hospital stays, mortality, and healthcare costs. Adequate nutrition is therefore crucial in the ICU. To ensure appropriate nutrition, accurate determination of total energy expenditure (TEE) is essential. In practice, predictive equations are often used, but these can misestimate TEE in ICU patients due to complex metabolic changes. Indirect calorimetry is recommended but limited by technical constraints. Consequently, the doubly labeled water (DLW) method, though expensive, offers a precise and non-invasive way to measure TEE over time.

This study applies the DLW method in ICU patients to improve energy assessment and guide personalized nutrition strategies that support recovery and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the ICU of Jessa Hospital
* Male and female sexes
* Age: > 18 years old
* Expected ICU stay of 5 days or more

Exclusion Criteria:

* Dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Energy expenditure | Min: 1-5 days; Max: 1-20 days
  Measured using the DLW method by only taking urine samples

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital Campus Virga Jesse, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No